CLINICAL TRIAL: NCT00726115
Title: Safety, Tolerability, and Pharmacokinetics, of Single and Multiple Dose of SAM-531 Administered Orally To Healthy Young and Elderly Subjects
Brief Title: Study Evaluating Safety, Tolerability and Pharmacokinetics of Single and Multiple Dose of SAM-531
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3193A1-1111
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-531

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): arm placebo
  Interventions: Drug: SAM-531
- 2 (Experimental): arm drug
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SAM-531
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
The main objectives of this study is to assess the safety and tolerability of ascending single and multiple oral doses of SAM-531 in healthy subjects

ELIGIBILITY:
Inclusion criteria:

* Body mass index in the range of 18 to 30 kg/m2 and body weight greater than or equal to 50 kg. Body weight for elderly subjects must be greater than or equal to 45 kg.
* history, physical examination findings, clinical laboratory test results, vital sign measurements, and digital 12-lead ECG readings.

Exclusion criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal (GI), endocrine, immunologic, dermatologic, hematologic, neurologic or psychiatric disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics, routine Lab tests, Vital signs, ECG | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Rueil-Malmaison, France